CLINICAL TRIAL: NCT01522989
Title: A Phase I Study of the CDK4/6 Inhibitor PD-0332991, 5-Fluorouracil, and Oxaliplatin in Patients With Advanced Solid Tumor Malignancies
Brief Title: PD-0332991, 5-FU, and Oxaliplatin for Advanced Solid Tumor Malignancies
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Georgetown University (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2011-219; WS1877559 (Other: Pfizer)
Record Dates: First submitted 2011-12-20; First posted 2012-02-01 (Estimated); Last update posted 2020-03-04 (Actual); Status verified 2019-05

CONDITIONS: Advanced Solid Tumor Malignancies
Keywords: Cancer; Advanced; Refractory
MeSH Terms: conditions — Neoplasms | interventions — palbociclib; Fluorouracil; Oxaliplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- PD-0332991, 5-FU and oxaliplatin (Experimental): PD-0332991 with 5-FU and oxaliplatin
  Interventions: Drug: PD-0332991; Drug: 5-FU; Drug: Oxaliplatin

INTERVENTIONS:
Drug: PD-0332991 — Stage 1:
  PD-0332991 daily Days 1-7 in escalating doses 5-FU 400 mg/m2 Day 8 Leucovorin 400 mg/M2 Day 8 5-FU continuous Infusion over 46 hours, 2400 mg/M2 Days 8-10
  Stage 2: 3 cohorts of subjects each will be treated with the dose of PD-0332991 determined to be the recommended Phase 2 dose in Stage 1 of the study with 5-FU at the doses above but on different schedules:
  Cohort 1: 5-FU bolus on Day 7 and infusion Days 7-9 Cohort 2: 5-FU bolus Day 9 and infusion Days 9-11 Cohort 3: 5-FU bolus Day 1 and infusion Days 1-3
  In Stage 3, PD-0332991 and 5-FU will be given at the doses and schedule determined in Stages 1 and 2 of this study with the addition of oxaliplatin 85 mg/m2 given on the same day as the 5-FU bolus.
  Other Names: Palbociclib
Drug: 5-FU — Stage 1:
  PD-0332991 daily Days 1-7 in escalating doses 5-FU 400 mg/m2 Day 8 Leucovorin 400 mg/M2 Day 8 5-FU continuous Infusion over 46 hours, 2400 mg/M2 Days 8-10
  Stage 2: 3 cohorts of subjects each will be treated with the dose of PD-0332991 determined to be the recommended Phase 2 dose in Stage 1 of the study with 5-FU at the doses above but on different schedules:
  Cohort 1: 5-FU bolus on Day 7 and infusion Days 7-9 Cohort 2: 5-FU bolus Day 9 and infusion Days 9-11 Cohort 3: 5-FU bolus Day 1 and infusion Days 1-3
  In Stage 3, PD-0332991 and 5-FU will be given at the doses and schedule determined in Stages 1 and 2 of this study with the addition of oxaliplatin 85 mg/m2 given on the same day as the 5-FU bolus.
  Other Names: 5-Fluorouracil
Drug: Oxaliplatin — Stage 1:
  PD-0332991 daily Days 1-7 in escalating doses 5-FU 400 mg/m2 Day 8 Leucovorin 400 mg/M2 Day 8 5-FU continuous Infusion over 46 hours, 2400 mg/M2 Days 8-10
  Stage 2: 3 cohorts of subjects each will be treated with the dose of PD-0332991 determined to be the recommended Phase 2 dose in Stage 1 of the study with 5-FU at the doses above but on different schedules:
  Cohort 1: 5-FU bolus on Day 7 and infusion Days 7-9 Cohort 2: 5-FU bolus Day 9 and infusion Days 9-11 Cohort 3: 5-FU bolus Day 1 and infusion Days 1-3
  In Stage 3, PD-0332991 and 5-FU will be given at the doses and schedule determined in Stages 1 and 2 of this study with the addition of oxaliplatin 85 mg/m2 given on the same day as the 5-FU bolus.
  Other Names: Eloxatin

SUMMARY:
This study is for patients with advanced solid tumor malignancies (cancer that has spread to other parts of the body).

The purpose of this study is to test the safety and effectiveness of a new combination of drugs, PD-0332991 and 5-Fluorouracil and Oxaliplatin for patients with advanced solid tumor malignancies . PD-0332991 stops cells from dividing by blocking an enzyme called cyclin-dependent kinase (CDK), which cancer cells need to grow and divide. By inhibiting this enzyme, PD-0332991 prevent cancer cells from growing and dividing, while the 5-Fluorouracil and Oxaliplatin damage the cells, hopefully increasing the killing of cancer cells, thus decreasing the tumors in the body.

PD-0332991 is an investigational or experimental anti-cancer agent that has not yet been approved by the Food and Drug Administration for use in colorectal cancer. It is given as a pill which is taken once a day for one week followed by one week off. 5-Fluorouracil and Oxaliplatin are administered as an infusion into a vein once every 2 weeks and are approved for and used as chemotherapy for several cancers.

ELIGIBILITY:
Inclusion Criteria:

* Retinoblastoma-positive, histologically proven advanced solid tumor malignancies for which no curative therapy exists
* Biopsy accessible tumor deposits
* Corrected QT interval less than 500 milliseconds by EKG
* ECOG preformance status 0-2
* Subjects with no brain metastases or a history of previously treated brain metastases who have been treated by surgery or stereotactic radiosurgery at least 4 weeks prior to enrollment and have a baseline MRI that shows no evidence of active intracranial disease and have not had treatment with steroids within 1 week of study enrollment.
* Adequate hepatic, bone marrow, and renal function
* Partial thromboplastin time must be </= 1.5 x upper limit normal range and INR < 1.5. Subjects on anticoagulant will be permitted to enroll as long as the INR is in acceptable therapeutic range.
* Life expectancy > 12 weeks
* Women of childbearing potential must have a negative serum pregnancy test within 14 days prior to initiation of treatment and/or postmenopausal women must be amenorrheic for at least 12 months.
* Subject is capable of understanding and complying with parameters of the protocol and able to sign and date the informed consent.

Exclusion Criteria:

* Intolerant of, or ineligible for 5-FU, oxaliplatin and/or the combination of both
* CNS metastases that do not meet the criteria outlined in the inclusion criteria
* Peripheral neuropathy >/= Grade 2 at baseline or peripheral neuropathy >/= Grade 1 with neuropathic pain
* Active severe infection or known chronic infection with HIV or hepatitis B virus
* Cardiovascular disease problems including unstable angina, therapy for life-threatening ventricular arrhythmia or myocardial infarction, stroke, or congestive heart failure within the last 6 months.
* Life-threatening visceral disease or other severe concurrent disease
* Women who are pregnant or breastfeeding
* Anticipated patient survival under 3 months
* Concurrent use of known CYP 3A4 inhibiting or activating medications
* Clinically significant and uncontrolled major medical condition(s)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2011-12; Primary Completion 2020-12 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Recommended Phase 2 dose and schedule | 18 months
  The dose and schedule of PD-0332991 to be used in combination with 5-FU

SECONDARY OUTCOMES:
Toxicity of the combination of PD-0332991, 5-FU, and oxaliplatin | 18 months
  To quantify the adverse events
Pharmacodynamics | 18 months
  evaluation of the effects of schedule of therapy on pharmacodynamic measures of PD-0332991 activity
Response rate | 18 months
  Response rate as determined by RECIST 1.1
Disease control rate | 4 months
  Stable disease after four cycles + partial response + complete response
Trough level of PD-0332991 on Day 1 of Cycles 1-4 | 4 months
  Determination of the effects of 5-FU on pharmacokinetics of PD-0332991

CONTACTS AND LOCATIONS:
Overall Officials: Michael Pishvaian, MD PhD, Principal Investigator — Georgetown University
Locations (1):
- Georgetown Lombardi Comprehensive Cancer Center, Washington D.C., District of Columbia, United States